CLINICAL TRIAL: NCT03021096
Title: Natural History of Pain After Shoulder Arthroplasty Conducted With Multimodal Analgesia
Acronym: TSA
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0779
Record Dates: First submitted 2017-01-03; First posted 2017-01-13 (Estimated); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-01

CONDITIONS: TSA; Bruise; Pain, Postoperative
MeSH Terms: conditions — Contusions; Pain, Postoperative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Surveys — The study is just using validated surveys to assess pain and mood states after surgery

SUMMARY:
This study aims to identify the timeline of pain following total shoulder replacement with the goal of developing data for a subsequent randomized trial. The investigators believe that with using HSS's current protocol, many patients have postoperative pain that is no worse than their preoperative pain. Previous HSS anesthesia protocols for total shoulder arthroplasty patients have not formally followed patients past their hospital discharge, and the investigators believe that some patients do experience moderate to severe subacute postoperative pain. Therefore, this study's primary outcome is to look at the numeric pain scores at 14 days after surgery. Future studies will look at measures of preventing bruising and subsequent pain after shoulder replacement.

DETAILED DESCRIPTION:
This is a pilot study, with the goals of

1. developing data for a subsequent randomized trials
2. describing the pain trajectory after total shoulder arthroplasty given comprehensive multimodal perioperative analgesia
3. gathering preliminary data about which shoulder arthroplasty patients are at high risk for moderate or severe postoperative pain (NRS with movement, POD14, moderate >= 4- 6; Gerbershagen 2011; severe >= 7-10, Krebs 2007) Potential factors include fibromyalgia score, catastrophizing score, anxiety/depression score, gender, preoperative opioid use
4. gathering preliminary data on the potential association between the predictors listed in (c) and NRS pain score with movement on POD 14.
5. estimating incidence and severity of postoperative bruising on POD 14

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for the standardized anesthetic for TSA
* Patients who are capable to provide informed consent and answer questions in English (Study involves questionnaires validated in English)
* Age 18-80

Exclusion Criteria:

* Incapable to provide informed consent
* Contraindications for regional anesthesia (anticoagulation, infection at injection site)
* Patients undergoing TSA for Trauma or Rheumatoid Arthritis
* Revision TSA (previous non-TSA surgery is not an exclusion)
* Conversion of hemiarthroplasty to TSA
* Planned use of tranexamic acid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing TSA for Osteoarthritis, Reverse, Anatomic procedures
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques YaDeau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Goon AK, Dines DM, Craig EV, Gordon MA, Goytizolo EA, Lin Y, Lin E, YaDeau JT. A clinical pathway for total shoulder arthroplasty-a pilot study. HSS J. 2014 Jul;10(2):100-6. doi: 10.1007/s11420-014-9381-0. Epub 2014 Mar 8. PMID 25050091
- [Background] YaDeau JT, Gordon MA, Goytizolo EA, Lin Y, Fields KG, Goon AK, Holck G, Miu TW, Gulotta LV, Dines DM, Craig EV. Buprenorphine, Clonidine, Dexamethasone, and Ropivacaine for Interscalene Nerve Blockade: A Prospective, Randomized, Blinded, Ropivacaine Dose-Response Study. Pain Med. 2016 May;17(5):940-60. doi: 10.1093/pm/pnv010. Epub 2015 Dec 14. PMID 26814246

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Shoulder Surgery Patients: In the operating room, patients received intravenous sedation of up to 5 mg of midazolam, 10 to 20 mg of ketamine, and propofol as deemed appropriate. An ultrasound-guided interscalene peripheral nerve block was performed in the operating room, before surgery, using 25 mL bupivacaine, 0.5%, with added 100 mg clonidine, 2 mg preservative free dexamethasone, and 150 mg buprenorphine. During the procedure, patients received either intravenous sedation with a propofol infusion, or general anesthesia with propofol induction, either laryngeal mask airway or endotracheal tube insertion, and general anesthesia maintenance with titrated propofol and 1% sevoflurane. For the intravenous sedation and general anesthesia groups, patients received ketamine (total of 50 mg), ondansetron (4 mg), famotidine (20 mg), dexamethasone (4 mg) and ketorolac (15 mg) during surgery. For postoperative analgesia, patients received intravenous acetaminophen (1000 mg every 6 hours, four total doses) and intravenous ketorolac (15 mg every 8 hours, for three postoperative doses in addition to one dose in the operating room) followed by oral acetaminophen (650 mg every 6 hours for 3 days) and oral meloxicam (7.5-15 mg per day). Oral opioids were available on demand, based on patient description of pain to the nursing staff as mild, moderate, or severe. Each patient also received intravenous patient-controlled analgesia of hydromorphone.
Period: Overall Study
Arm/Group | Total Shoulder Surgery Patients
Started | 108
Completed | 102
Not Completed | 6
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale Pain Scores at Post-operative Day 14
Description: Quantifying patients' pain at a sub-acute time point after surgery at rest and with movement.
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Time Frame: 14 days after surgery for each patient
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
score on a scale
  NRS at rest | 1.6 (1.8)
  NRS with movement | 3.1 (2.3)

2. Secondary Outcome: Numeric Rating Scale (NRS) Pain With Movement and at Rest.
Description: The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". A lower score is a better outcome.
Time Frame: Days 1 day (POD0), 3 days(POD3), 7 days(POD7) and 3 months(POD90) after surgery
Population: some patients did not fill out questionnaire or were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
score on a scale
  NRS POD1 at rest: number analyzed (Participants) | 101
  NRS POD1 at rest | 1.6 (2.1)
  NRS POD1 with movement: number analyzed (Participants) | 43
  NRS POD1 with movement | 2.7 (3)
  NRS POD3 at rest: number analyzed (Participants) | 95
  NRS POD3 at rest | 2.8 (3.3)
  NRS POD3 with movement: number analyzed (Participants) | 83
  NRS POD3 with movement | 4.7 (2.4)
  NRS POD7 at rest: number analyzed (Participants) | 88
  NRS POD7 at rest | 2.3 (2.4)
  NRS POD7 with movement: number analyzed (Participants) | 86
  NRS POD7 with movement | 3.9 (2.3)
  NRS POD90 at rest: number analyzed (Participants) | 83
  NRS POD90 at rest | 0.8 (1.7)
  NRS POD90 with movement: number analyzed (Participants) | 83
  NRS POD90 with movement | 1.7 (2.2)

3. Secondary Outcome: Opioid Consumption (in Past 24 Hours)
Description: Measured in milligrams taken. A lower consumption is a better outcome.
Time Frame: Days 1 day, 3 days, 7 days after surgery
Population: some patients were lost to follow up.
Measure: Median (Inter-Quartile Range); unit: oral morphine equivalents (mg)
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
oral morphine equivalents (mg)
  POD1 | 17.5 [3.9 to 50.1]
  POD3 | 30 [7.4 to 63.2]
  POD7 | 10 [0 to 37.5]

4. Secondary Outcome: Opioid Related Symptom Distress Scale
Description: The Opioid-Related Symptom Distress Scale (ORSDS) is calculated by taking the average of the three symptom distress dimensions. Frequency will be assessed using a 4 point scale: 1, rarely 2, occasionally 3, frequently 4, almost constantly with 1 being the lowest and 4 being the highest. Severity is assessed using a 4 point scale: 1, slight 2, moderate 3, severe 4, very severe with 1 being the lowest and 4 being the highest. Bothersomeness is assessed using a 5 point scale: 1, not at all 2, a little bit 3, somewhat 4, quite a bit 5, very much with 1 being the lowest and 5 being the highest.
  A higher score indicates worse outcomes. The total score for each participant is calculated and the median score for all participants is reported.
Time Frame: Day 1 after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
score on a scale | 0.3 [0.1 to 0.5]

5. Secondary Outcome: Range of Motion
Description: Measure the ability of shoulder movement from 0 to 180 degrees at these follow up visits with the surgeon after surgery.
Time Frame: Day 14 after surgery and 3 months after surgery
Population: some patients were lost to follow up or did not answer questionnaire.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
degrees
  14 days after surgery extension: number analyzed (Participants) | 26
  14 days after surgery extension | 15.8 (5.8)
  3 months after surgery extension: number analyzed (Participants) | 2
  3 months after surgery extension | 35 (21.2)

6. Secondary Outcome: Severity of Bruising
Description: Surgeon will assess each individual patient to determine whether bruising occurred and if so, the size and severity of the bruise.
Time Frame: Day 14 after surgery
Population: some patients were lost to follow up or did not complete questionnaire. 32 people were reported to have bruising and size (in centimeters) of their bruises were measured.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 32
cm | 1.5 (1.9)

7. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: The Hospital Anxiety and Depression Scale (HADS) measures anxiety and depression in a general medical population of patients. a lower score is a better outcome. Each item on the questionnaire is scored from 0-3 and a person's total score can ranged from 0 = normal and 21 = abnormal for either anxiety or depression.
  Scale range:
  0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
  A total score for each participant was calculated and then all participants' scores were averaged.
Time Frame: Day 1 after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
score on a scale
  Anxiety | 4.1 (3.3)
  Depression | 3.9 (2.7)

8. Secondary Outcome: PainOUT Questionnaire
Description: The PainOUT questionnaire assess pain intensity, quality of pain, and satisfaction with pain management. The questionnaire measured the following:
  1. Worst pain: On a 0-10 scale, where 0 means "no pain" and 10 means "worst possible pain". Higher scores reflect more severity.
  2. Pain severity: On a scale 0-10, where 0 means "very unsatisfied" and 10 means "very satisfied". Higher scores means more satisfaction.
  3. Interference with sleep: Rated on a 0-10 scale, where 0 means "does not interfere" and 10 means "completely interfere" A higher rating means more interference.
  4. Nausea & Itching: Both rated on a 0-10 scale, where 0 means "none" and 10 means "severe". A higher rating means more severe.
  5. Drowsiness: Rated on a 0-10 scale, where 0 means "not at all" and 10 means "extremely". A higher rating means more severe.
  Each question score for each participant was added up and divided by the total number of participants to obtain an average score of 0-10 at each timepoint.
Time Frame: Day 1 and 14 after surgery
Population: some patients were lost to follow up.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
score on a scale
  POD1 - Worst pain: number analyzed (Participants) | 97
  POD1 - Worst pain | 2 [0 to 5]
  POD14 - Worst pain: number analyzed (Participants) | 94
  POD14 - Worst pain | 4 [2 to 6]
  POD1 - Pain severity | 0 [0 to 0]
  POD14 - Pain severity | 0 [0 to 10]
  POD1 - Interference with sleep | 0 [0 to 2]
  POD14 - Interference with sleep | 0 [0 to 5]
  POD1 - Nausea | 0 [0 to 0]
  POD14 - Nausea | 0 [0 to 0]
  POD1 - Itching | 0 [0 to 0]
  POD14 - Itching | 0 [0 to 1]
  POD1 - Drowsiness | 0 [0 to 5]
  POD14 - Drowsiness | 0 [0 to 2]

9. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The pain catastrophizing scale (PCS) evaluates a person's pain experience by asking them how they feel and what they think about when they are in pain.
  The questionnaire uses a 5-point Likert scale, with answers ranging from 0 (never) to 4. (always). The total score is the sum of the individual item scores and ranges from 0 to 52. A lower score indicates a more positive outcome.
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
score on a scale | 12 (11.9)

10. Secondary Outcome: Fibromyalgia Scale. a Lower Score is a Better Outcome.
Description: The symptom severity (SS) scale assesses four symptoms that are thought to be defining in a fibromyalgia diagnosis.
  The four symptoms assessed by the criteria are as follows:
  1. Fatigue
  2. Waking from sleep feeling unrefreshed
  3. Cognitive symptoms (including trouble concentrating, confusion, disorientation, and impaired comprehension)
  4. Somatic symptoms (physical sensations such as pain, dizziness, nausea, fainting, or bowel disorders)
  Each of the 4 symptoms is graded on a scale of 0 to 3, with 0 indicating no symptoms, 1 indicating mild symptoms, 2 indicating moderate symptoms, and 3 indicating severe symptoms. The sum of the scores for each of the 4 symptoms is summed to produce the SS total score. The SS total score has a minimum score of 0 and a maximum score of 12.
  The higher score means worst outcome. The sum score for each participant is calculated and then the average score for all participants is reported.
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Shoulder Surgery Patients
Number analyzed (Participants) | 102
score on a scale | 5.5 (3.4)

ADVERSE EVENTS:
Time Frame: 3 months after surgery
Arm/Group | Total Shoulder Surgery Patients
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT03021096/Prot_SAP_000.pdf